CLINICAL TRIAL: NCT06771141
Title: The Impact of Virtual Reality Application Before Endoscopy on Anxiety and Vital Signs in Children
Brief Title: Virtual Reality Before Pediatric Endoscopy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yuzuncu Yil University (Other)
Responsible Party: Principal Investigator, mehmet bulduk, PhD, Yuzuncu Yil University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2024/07-25
Record Dates: First submitted 2025-01-08; First posted 2025-01-13 (Actual); Last update posted 2025-01-14 (Actual); Status verified 2024-07

CONDITIONS: Pediatric Anxiety Disorders
Keywords: Virtual Reality, Anxiety, Endoscopy, Pediatric, Vital Signs
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: his study uses a randomized controlled trial (RCT) design with a parallel assignment model. Participants are divided into two groups: the intervention group, which receives a virtual reality (VR) application before undergoing endoscopy, and the control group, which receives standard care. The study is open-label, meaning both participants and researchers are aware of the group assignments. This design allows for a direct comparison of the effects of the VR application on anxiety levels and vital signs in pediatric patients.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Virtual Reality Intervention Group (Experimental): This arm includes participants who will receive a 10-minute virtual reality (VR) session before their endoscopy procedure. The VR intervention aims to reduce anxiety and stabilize vital signs (e.g., systolic/diastolic blood pressure, heart rate, oxygen saturation) by providing an immersive and interactive experience designed to distract and relax the participants. Anxiety levels and vital signs will be measured pre- and post-intervention to evaluate its effectiveness.
  Interventions: Behavioral: Virtual Reality Video Session
- Standard Care Control Group (No Intervention): Participants in this group will receive standard care prior to the endoscopy procedure, without the VR intervention. Anxiety levels and vital signs will be measured at similar intervals to compare with the experimental group.

INTERVENTIONS:
Behavioral: Virtual Reality Video Session — This intervention involves a 10-minute virtual reality (VR) video session designed to reduce pre-procedural anxiety and promote relaxation in pediatric patients. The video immerses participants in a calming virtual environment with interactive and visually engaging content tailored for children. It is administered prior to the endoscopy procedure to help manage anxiety and stabilize vital signs, such as blood pressure, heart rate, and oxygen saturation. The VR session serves as a non-pharmacological approach to anxiety management during medical procedures.
  Arms: Virtual Reality Intervention Group

SUMMARY:
Brief Summary: Clinical Study

The purpose of this clinical study is to evaluate whether the use of virtual reality (VR) before endoscopy reduces anxiety levels and positively impacts vital signs in children. This study aims to answer the following key questions:

Does the VR application reduce pre-endoscopy anxiety in children? Does the VR application improve vital signs such as heart rate, blood pressure, and oxygen saturation in children?

Researchers will compare the effects of the VR application with standard care to assess its effectiveness.

Participants:

The experimental group will undergo a 15-minute VR session before the endoscopy.

The control group will receive standard care without VR. Anxiety levels and vital signs will be measured throughout the study.

This study aims to explore whether VR technology can serve as an effective stress management tool during pediatric medical procedure

ELIGIBILITY:
Inclusion Criteria:

* Children aged 8 to 17 years.
* Scheduled to undergo an endoscopy procedure.
* Able to provide assent, and their parents or legal guardians provide written informed consent.
* No prior exposure to virtual reality applications.
* Willing to participate in the study.

Exclusion Criteria:

* Presence of a chronic medical condition affecting cardiovascular or respiratory systems.
* Diagnosed with a severe psychiatric disorder.
* Known visual or auditory impairments that could prevent participation in a virtual reality session.
* History of seizures or epilepsy.
* Unwillingness to participate or inability to comply with study procedures.

Ages: 8 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 80 (Actual)
Dates: Start 2024-07-29 (Actual); Primary Completion 2024-11-26 (Actual); Study Completion 2024-12-15 (Actual)

PRIMARY OUTCOMES:
Reduction in Anxiety Levels in Pediatric Patients | Anxiety levels will be measured immediately before the intervention and immediately after the intervention on the same day as the endoscopy procedure.
  The primary outcome measure is the change in anxiety levels among pediatric patients undergoing endoscopy. Anxiety levels will be assessed using the State-Trait Anxiety Inventory for Children (STAIC), a validated tool for measuring anxiety in children. Scores will be measured before and after the intervention to determine the effectiveness of the virtual reality (VR) application compared to the control group receiving standard care.

CONTACTS AND LOCATIONS:
Locations (1):
- Van Yüzüncü Yıl Üniversity, Van, Van, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Individual Participant Data (IPD) will not be shared to prioritize the privacy and confidentiality of participants. Additionally, it has been specified in the ethical approval that the data will only be used for the purposes of this study and will not be shared with third parties.